CLINICAL TRIAL: NCT02367352
Title: A Phase 1b Study of Alisertib (MLN8237) in Combination With Weekly Paclitaxel in East Asian Patients With Advanced Solid Tumors
Brief Title: Alisertib (MLN8237) in Combination With Weekly Paclitaxel in East Asian Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C14022; U1111-1164-7696 (Registry Identifier: WHO); JapicCTI-152845 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2015-02-11; First posted 2015-02-20 (Estimated); Results first posted 2019-05-02 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Advanced Solid Tumors; Ovarian Cancer; Small Cell Lung Cancer
Keywords: Drug therapy; Dose escalation; Dose expansion
MeSH Terms: conditions — Ovarian Neoplasms; Small Cell Lung Carcinoma | interventions — MLN 8237; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Dose Escalation Phase) (Experimental): Alisertib 15 mg, tablet, orally, twice daily, (3 days on/4 days off for 3 weeks) on Days 1 to 3, 8 to 10 and 15 to 17 in 28 day cycles in combination with Paclitaxel 60 mg/m^2, intravenous (IV), on Days 1, 8, and 15 in a 28-day cycle until disease progression or unacceptable toxicity (Up to 22 Cycles).
  Interventions: Drug: Alisertib; Drug: Paclitaxel
- Cohort 2 (Dose Escalation Phase) (Experimental): Alisertib 25 mg, tablet, orally, twice daily, (3 days on/4 days off for 3 weeks) on Days 1 to 3, 8 to 10 and 15 to 17 in 28 day cycles in combination with Paclitaxel 60 mg/m^2, intravenous (IV), on Days 1, 8, and 15 in 28-day cycle until disease progression or unacceptable toxicity. Dose of alisertib will be de-escalated to 20 mg if ≥ 2 participants experience a dose limiting toxicity (DLT).
  Interventions: Drug: Alisertib; Drug: Paclitaxel
- Dose Expansion Cohort (Experimental): Alisertib, MTD/RP2D determined in Dose Escalation Phase, orally, twice daily, (3 days on/4 days off for 3 weeks) on Days 1 to 3, 8 to 10 and 15 to 17 in 28 day cycles in combination with Paclitaxel 60 mg/m^2, IV on Days 1, 8, and 15 in 28-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Alisertib; Drug: Paclitaxel

INTERVENTIONS:
Drug: Alisertib — Alisertib tablets
Drug: Paclitaxel — Paclitaxel intravenous solution

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability and determine the MTD to subsequently define an RP2D of alisertib in combination with weekly paclitaxel in East Asian participants with advanced solid tumors.

DETAILED DESCRIPTION:
The drug being tested in this study was called alisertib. Alisertib in combination with paclitaxel was tested to find a safe and well-tolerated dose in East Asian participants. The study consisted of 2 parts: a dose escalation phase to determine the maximum tolerated dose (MTD) and define the recommended phase 2 dose (RP2D) of the alisertib plus paclitaxel combination in East Asian participants with advanced solid tumors; the second part is an expansion cohort at the RP2D of the alisertib plus paclitaxel in East Asian participants with either ovarian cancer or small cell lung cancer. This study looked at safety (lab results and side effects) and pharmacokinetic properties (how the drugs move throughout the body).

This open label study enrolled 9 participants. Dose Escalation Phase: Alisertib tablets at a starting dose of 15 mg, orally, twice daily, 3 days on/4 days off for 3 weeks in 28 day cycle in combination with paclitaxel, 60 mg/m^2 intravenous on days 1, 8, and 15 in 28-day cycles in Cohort 1 escalated to a dose of 25 mg alisertib, orally, twice daily 3 days on/4 days off for 3 weeks in 28 day cycles in Cohort 2. If ≥ 2 participants experience a dose limiting toxicity (DLT) the dose of alisertib decreased to 20 mg. Expansion Cohort: alisertib tablets at the determined RP2D dose orally, twice daily 3 days on/4 days off for 3 weeks in 28 day cycles in combination with paclitaxel, 60 mg/m^2 intravenous. Treatment was continued until disease progression or unacceptable toxicity.

* Alisertib 15 mg to 25 mg tablets
* Paclitaxel 60 mg/m^2 intravenous solution

This multi-centre trial was conducted in Japan and Korea. The overall time to participate in this study was up to 24 months.

The study was terminated early because of the sponsor's decision. Enrollment was completed in the dose escalation cohort, but no participants were enrolled in the dose expansion cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants 18 years or older (or minimum age of legal consent consistent with local regulations) at the time written study informed consent is obtained.
2. Participants of East Asian ethnicity (eg, Chinese, Japanese, or Korean).
3. Must have a diagnosis of a solid tumor malignancy (escalation part) or relapsed or refractory ovarian cancer (OC) or small cell lung cancer (SCLC) (expansion part).

   * Participants in the expansion cohort must have a pathologically (histology or cytology) confirmed diagnosis of either OC (including recurrent epithelial ovarian, fallopian tube, or primary peritoneal cancer) or SCLC, which is measurable disease as per Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1.
   * Participants in the expansion cohort must not have received more than 2 prior taxane containing regimens.
4. No antineoplastic therapy (eg, drugs, biologicals, monoclonal antibodies, etc) or radiotherapy within the 3 weeks before enrollment (14 days for regimens with recovery expected within 7 to 14 days). The participant must have recovered (ie, ≤ Grade 1 toxicity or participant's baseline status, except alopecia) from all treatment-related toxicities.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Adequate bone marrow function as defined by:

   * Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3 (without need for growth factor support).
   * Platelet count ≥ 100,000 cells/mm3 (without need for transfusion or growth factor support).
   * Hemoglobin level ≥ 9 g/dL.
7. Adequate liver function as defined by:

   * Bilirubin < 1.5 times the upper limit of normal (ULN)
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN (≤ 5 x ULN if due to liver metastases)
   * Serum albumin equal to or greater than the lower limit of normal
8. Adequate renal function as defined by:

   * Creatinine clearance ≥ 30 mL/minute (can be calculated using serum creatinine value).
9. No more than 2 previous chemotherapy regimen in the metastatic setting.
10. Female participants who:

    * Are postmenopausal for at least 1 year before the screening visit, OR
    * Are surgically sterile, OR
    * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 30 days after the last dose of study drug
    * Adhere to any treatment-specific pregnancy prevention guidelines for paclitaxel

    Male participants, even if surgically sterilized (ie, status postvasectomy), who:
    * Agree to practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug
    * Adhere to any treatment-specific pregnancy prevention guidelines for paclitaxel.
11. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the participant at any time without prejudice to future medical care.
12. Suitable venous access for the study-required blood sampling, including pharmacokinetics (PK).
13. Ability to swallow tablets.

Exclusion Criteria:

1. Participants with carcinomatous meningitis.
2. Participants with symptomatic and/or progressive brain metastases or treatment with brain edema.
3. Known hypersensitivity to Cremophor® EL, paclitaxel, alisertib or their components.
4. Prior treatment with an Aurora A specific-targeted or pan-Aurora-targeted agent, including alisertib in any setting.
5. Prior history of ≥ Grade 2 neurotoxicity or any toxicity requiring discontinuation from taxane chemotherapy that is not resolved to ≤ Grade 1.
6. Participants who received prior weekly taxane-based therapy with early disease progression during or within 1 month of completing therapy (refractory disease).
7. Any comorbid condition or unresolved toxicity that would preclude administration of weekly paclitaxel.
8. Systemic treatment with moderate or strong CYP3A inhibitors must be discontinued at least 14 days before the first dose of alisertib, and the use of these agents is not permitted during the study.
9. Known gastrointestinal (GI) abnormality (including recurrent nausea or vomiting) or GI procedure that could interfere with or modify the oral intake, absorption, or tolerance of alisertib.
10. Participants requiring treatment with clinically significant enzyme inducers, such as the enzyme-inducing antiepileptic drugs phenytoin, carbamazepine, phenobarbital, oxcarbazepine, primidone, rifampin, rifabutin, rifapentine, or St. John's wort within 14 days before the first dose of alisertib or requiring the use of these medications during the study.
11. Requirement for administration of proton pump inhibitor (PPI), H2 antagonist (premedication for paclitaxel allowed), or pancreatic enzymes. Use of any PPI in either continued or intermittent use will be prohibited during the conduct of the study and participants must discontinue any use of PPI within 4 days before the first dose of alisertib.
12. Life-threatening or severe central nervous system (CNS), pulmonary, renal, or hepatic disease unrelated to cancer, or any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
13. Treatment with any investigational products within 5 half-lives before the first dose of study drug.
14. Treatment with fully human or chimeric monoclonal antibodies within 42 days before the first dose of study drug (21 days if clear evidence of progression).
15. Major surgery within 14 days before the first dose of study drug.
16. Infection requiring systemic intravenous (IV) antibiotic therapy within 14 days preceding the first dose of study drug, or other severe infection.
17. Known human immunodeficiency virus (HIV) positive.
18. Ongoing or active hepatitis B or hepatitis C infection. Testing is not required in the absence of clinical findings or suspicion.
19. History of myocardial infarction, unstable symptomatic ischemic heart disease, uncontrolled hypertension despite appropriate medical therapy, any ongoing cardiac arrhythmias of > Grade 2, thromboembolic events (eg, deep vein thrombosis, pulmonary embolism, or symptomatic cerebrovascular events), or any other cardiac condition (eg, pericardial effusion or restrictive cardiomyopathy) within 6 months before receiving the first dose of study drug. Chronic stable atrial fibrillation on stable anticoagulant therapy is allowed. Participants with a pacemaker may be enrolled in the study upon discussion with the project clinician.
20. Female participants who are in the lactation period or have a positive serum pregnancy test during the Screening period or a positive urine pregnancy test on Day1 before the first dose of study drug.
21. Diagnosed with or treated for another malignancy within 3 years before the first dose of study drug, or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with non-melanoma skin cancer or carcinoma in situ of any type may be enrolled in the study if they have undergone complete resection and no evidence of active disease is present.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-03-19 (Actual); Primary Completion 2017-05-23 (Actual); Study Completion 2017-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Millennium Pharmaceuticals, Inc.
Locations (3):
- Japan (2):
  - Chiba
  - Shizuoka
- Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 3 investigative sites in Japan and Republic of Korea from 19 March 2015 to 23 May 2017.
Pre-assignment Details: Participants with a diagnosis of Advanced Solid Tumors were enrolled in a dose escalation phase to receive a starting dose of alisertib 15 mg plus paclitaxel 60 mg/m^2. The dose expansion phase was not conducted.
Period: Overall Study
Arm/Group | Cohort 1 (Dose Escalation Phase) | Cohort 2 (Dose Escalation Phase) | Dose Expansion Cohort
Started | 9 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 9 | 0 | 0
Not completed — Progressive disease | 7 | 0 | 0
Not completed — Participant Received Alternative Therapy | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population is defined as all participants who received at least 1 dose of alisertib. Participants were only enrolled in Dose Escalation Cohort 1.
Arm/Group | Cohort 1 (Dose Escalation Phase)
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.48 (14.621)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 7
  Not reported | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 9
Region of Enrollment [Number; unit: participants]
  Japan | 3
  Korea, Republic Of | 6
Height [Mean (Standard Deviation); unit: cm] | 162.77 (6.907)
Weight [Mean (Standard Deviation); unit: kg] | 63.70 (10.165)
Body Surface Area [Mean (Standard Deviation); unit: m^2] | 1.693 (0.1542)

OUTCOME MEASURES:

1. Primary Outcome: Dose Escalation Phase: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. Preexisting conditions that worsened during the study were reported as adverse events.
  A SAE is any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.
Time Frame: From Day 1 to 30 days after the last dose of study drug (approximately 21 months)
Population: Safety population is defined as all participants who received at least 1 dose of alisertib. No participants were enrolled in Dose Escalation Phase Cohort 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Dose Escalation Phase) | Cohort 2 (Dose Escalation Phase)
Number analyzed (Participants) | 9 | 0
Participants
  AEs | 9 |
  SAEs | 4 |

2. Primary Outcome: Dose Escalation Phase: Number of Participants With Clinically Significant Laboratory Findings
Description: The number of participants with any markedly abnormal standard safety laboratory values including serum chemistry, hematology, and urine analysis will be collected throughout study. Laboratory values assessed by the investigator to be clinically significant were reported as adverse events.
Time Frame: From Day 1 to 30 days after the last dose of study drug (approximately 21 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Dose Escalation Phase) | Cohort 2 (Dose Escalation Phase)
Number analyzed (Participants) | 9 | 0
Participants
  Neutrophil Count Decreased | 5 |
  White Blood Cell Count Decreased | 4 |
  Blood Antidiuretic Hormone Abnormal | 1 |

3. Primary Outcome: Dose Escalation Phase: Number of Participants With Clinically Significant Vital Sign Findings
Description: The number of participants with any markedly abnormal vital sign values (blood pressure, heart rate, and temperature) will be collected throughout study. Vital signs assessed by the investigator to be clinically significant were reported as adverse events.
Time Frame: From Day 1 to 30 days after the last dose of study drug (approximately 21 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Dose Escalation Phase) | Cohort 2 (Dose Escalation Phase)
Number analyzed (Participants) | 9 | 0
Participants | 1 |

4. Primary Outcome: Dose Escalation Phase: Cmax: Maximum Observed Plasma Concentration of Alisertib
Time Frame: Day 1 and Day 3 predose and at multiple time points (up to 12 hours) post-dose
Population: Pharmacokinetic data was not available as 9 participants were insufficient sample size to run the analysis.
Arm/Group | Cohort 1 (Dose Escalation Phase) | Cohort 2 (Dose Escalation Phase)
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Dose Escalation Phase: Tmax: Time to Reach the Maximum Plasma Concentration of Alisertib
Time Frame: Day 1 and Day 3 predose and at multiple time points (up to 12 hours) post-dose
Population: Pharmacokinetic data was not available as 9 participants were insufficient sample size to run the analysis.
Arm/Group | Cohort 1 (Dose Escalation Phase) | Cohort 2 (Dose Escalation Phase)
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Dose Escalation Phase: AUC(0-tau): Area Under the Plasma Concentration-time Curve From Time 0 to Time Tau Over the Dosing Interval for Alisertib
Time Frame: Day 1 and Day 3 predose and at multiple time points (up to 12 hours) post-dose
Population: Pharmacokinetic data was not available as 9 participants were insufficient sample size to run the analysis.
Arm/Group | Cohort 1 (Dose Escalation Phase) | Cohort 2 (Dose Escalation Phase)
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Dose Escalation Phase: Cmax: Maximum Observed Plasma Concentration of Paclitaxel
Time Frame: Day 1 predose and Day 1, 2 and 3 at multiple time points (up to 12 hours) post-dose
Population: Pharmacokinetic data was not available as 9 participants were insufficient sample size to run the analysis.
Arm/Group | Cohort 1 (Dose Escalation Phase) | Cohort 2 (Dose Escalation Phase)
Number analyzed (Participants) | 0 | 0

8. Primary Outcome: Dose Escalation Phase: Tmax: Time to Reach the Maximum Plasma Concentration of Paclitaxel
Time Frame: Day 1 predose and Day 1, 2, and 3 at multiple time points (up to 12 hours) post-dose
Population: Pharmacokinetic data was not available as 9 participants were insufficient sample size to run the analysis.
Arm/Group | Cohort 1 (Dose Escalation Phase) | Cohort 2 (Dose Escalation Phase)
Number analyzed (Participants) | 0 | 0

9. Primary Outcome: Dose Escalation Phase: AUC(0-tlast): Area Under the Plasma Concentration Curve From Time Zero to the Time of the Last Quantifiable Concentration of Paclitaxel
Time Frame: Day 1 predose and Day 1, 2, and 3 at multiple time points (up to 12 hours) post-dose
Population: Pharmacokinetic data was not available as 9 participants were insufficient sample size to run the analysis.
Arm/Group | Cohort 1 (Dose Escalation Phase) | Cohort 2 (Dose Escalation Phase)
Number analyzed (Participants) | 0 | 0

10. Primary Outcome: Dose Escalation Phase: AUC(0-inf): Area Under the Plasma Concentration-Time Curve From Tme 0 to Infinity
Time Frame: Day 1 predose and Day 1, 2, and 3 at multiple time points (up to 12 hours) post-dose
Population: Pharmacokinetic data was not available as 9 participants were insufficient sample size to run the analysis.
Arm/Group | Cohort 1 (Dose Escalation Phase) | Cohort 2 (Dose Escalation Phase)
Number analyzed (Participants) | 0 | 0

11. Primary Outcome: Dose Escalation Phase: T½: Terminal Phase Elimination Half-Life of Paclitaxel
Time Frame: Day 1 predose and Day 1, 2, and 3 at multiple time points (up to 12 hours) post-dose
Population: Pharmacokinetic data was not available as 9 participants were insufficient sample size to run the analysis.
Arm/Group | Cohort 1 (Dose Escalation Phase) | Cohort 2 (Dose Escalation Phase)
Number analyzed (Participants) | 0 | 0

12. Primary Outcome: Dose Expansion Phase: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: as for outcome 1
Time Frame: From Day 1 to 30 days after the last dose of study drug
Population: The dose expansion phase was cancelled by the sponsor.
Arm/Group | Dose Expansion Cohort
Number analyzed (Participants) | 0

13. Primary Outcome: Dose Expansion Phase: Number of Participants With Clinically Significant Laboratory Findings
Description: The number of participants with any markedly abnormal standard safety laboratory values will be collected throughout study.
Time Frame: From Day 1 to 30 days after the last dose of study drug
Population: The dose expansion phase was cancelled by the sponsor.
Arm/Group | Dose Expansion Cohort
Number analyzed (Participants) | 0

14. Primary Outcome: Dose Expansion Phase: Number of Participants With Clinically Significant Vital Sign Findings
Description: The number of participants with any markedly abnormal vital sign values will be collected throughout study.
Time Frame: From Day 1 to 30 days after the last dose of study drug
Population: The dose expansion phase was cancelled by the sponsor.
Arm/Group | Dose Expansion Cohort
Number analyzed (Participants) | 0

15. Primary Outcome: Dose Expansion Phase: Cmax: Maximum Observed Plasma Concentration of Alisertib
Time Frame: Day 1 and Day 3 predose and at multiple time points (up to 12 hours) post-dose
Population: The dose expansion phase was cancelled by the sponsor.
Arm/Group | Dose Expansion Cohort
Number analyzed (Participants) | 0

16. Primary Outcome: Dose Expansion Phase: Tmax: Time to Reach the Maximum Plasma Concentration of Alisertib
Time Frame: Day 1 and Day 3 predose and at multiple time points (up to 12 hours) post-dose
Population: The dose expansion phase was cancelled by the sponsor.
Arm/Group | Dose Expansion Cohort
Number analyzed (Participants) | 0

17. Primary Outcome: Dose Expansion Phase: AUC(0-tau): Area Under the Plasma Concentration-time Curve From Time 0 to Time Tau Over the Dosing Interval for Alisertib
Time Frame: Day 1 and Day 3 predose and at multiple time points (up to 12 hours) post-dose
Population: The dose expansion phase was cancelled by the sponsor.
Arm/Group | Dose Expansion Cohort
Number analyzed (Participants) | 0

18. Primary Outcome: Dose Expansion Phase: Cmax: Maximum Observed Plasma Concentration of Paclitaxel
Time Frame: Day 1 predose and Day 1, 2, and 3 at multiple time points (up to 12 hours) post-dose
Population: The dose expansion phase was cancelled by the sponsor.
Arm/Group | Dose Expansion Cohort
Number analyzed (Participants) | 0

19. Primary Outcome: Dose Expansion Phase: Tmax: Time to Reach the Maximum Plasma Concentration of Paclitaxel
Time Frame: Day 1 predose and Day 1, 2, and 3 at multiple time points (up to 12 hours) post-dose
Population: The dose expansion phase was cancelled by the sponsor.
Arm/Group | Dose Expansion Cohort
Number analyzed (Participants) | 0

20. Primary Outcome: Dose Expansion Phase: AUC(0-tlast): Area Under the Plasma Concentration Curve From Time Zero to the Time of the Last Quantifiable Concentration of Paclitaxel
Time Frame: Day 1 predose and Day 1, 2, and 3 at multiple time points (up to 12 hours) post-dose
Population: The dose expansion phase was cancelled by the sponsor.
Arm/Group | Dose Expansion Cohort
Number analyzed (Participants) | 0

21. Primary Outcome: Dose Expansion Phase: AUC(0-inf): Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity of Paclitaxel
Time Frame: Day 1 predose and Day 1, 2, and 3 at multiple time points (up to 12 hours) post-dose
Population: The dose expansion phase was cancelled by the sponsor.
Arm/Group | Dose Expansion Cohort
Number analyzed (Participants) | 0

22. Primary Outcome: Dose Expansion Phase: T½: Terminal Phase Elimination Half-Life of Paclitaxel
Time Frame: Day 1 predose and Day 1, 2, and 3 at multiple time points (up to 12 hours) post-dose
Population: The dose expansion phase was cancelled by the sponsor.
Arm/Group | Dose Expansion Cohort
Number analyzed (Participants) | 0

23. Secondary Outcome: Dose Expansion Phase: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants with complete response (CR) and partial response (PR) according to disease response based on the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Time Frame: Day 21 of every other Cycle beginning with Cycle 2 (Up to 12 months)
Population: The dose expansion phase was cancelled by the sponsor.
Arm/Group | Dose Expansion Cohort
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: First dose of study drug through 30 days after the last dose of any study drug (approximately 21 months)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Participants were only enrolled in Dose Escalation Cohort 1.
Arm/Group | Cohort 1 (Dose Escalation Phase)
All-Cause Mortality (participants affected / at risk) | 1/9
Serious Adverse Events (participants affected / at risk) | 4/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (Dose Escalation Phase) (N=9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 1
Pneumonia (Infections and infestations) | 1
Small cell lung cancer (disease progression) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — One treatment-emergent death occurred during treatment with alisertib and is not related.
Dizziness (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (Dose Escalation Phase) (N=9)
Diarrhoea (Gastrointestinal disorders) | 5
Stomatitis (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Intestinal perforation (Gastrointestinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Fatigue (General disorders) | 5
Asthenia (General disorders) | 2
Chest pain (General disorders) | 1
Chills (General disorders) | 1
Influenza like illness (General disorders) | 1
Malaise (General disorders) | 1
Pyrexia (General disorders) | 1
Neutrophil count decreased (Investigations) | 5
White blood cell count decreased (Investigations) | 4
Blood antidiuretic hormone abnormal (Investigations) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Hyponatraemia (Metabolism and nutrition disorders) | 3
Decreased appetite (Metabolism and nutrition disorders) | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 3
Bronchitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Delirium (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Dry eye (Eye disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Superior vena cava syndrome (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-01-25): https://cdn.clinicaltrials.gov/large-docs/52/NCT02367352/SAP_000.pdf
  • Study Protocol (2015-06-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT02367352/Prot_001.pdf